CLINICAL TRIAL: NCT00458354
Title: A Prospective, Multi-Center, Randomized Controlled Study to Compare the Spinal Sealant System as an Adjunct to Sutured Dural Repair With Standard of Care Methods During Spinal Surgery
Brief Title: Use of Spinal Sealant System During Spinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Confluent Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-0641
Record Dates: First submitted 2007-03-29; First posted 2007-04-10 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Spine Surgery; Excessive Repair; Spinal Cord Injuries; Complication of Surgical Procedure
Keywords: Spinal Sealant; Spinal Sealant System; Dural Repair; Spinal Surgery
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Sealant (Experimental): Dural repair with the Spinal Sealant System.
  Interventions: Device: Spinal Sealant
- Standard Methods (Active Comparator): Dural repair with standard methods such as the closing of the dura with stitches.
  Interventions: Procedure: Standard Methods of Closing of the Dura

INTERVENTIONS:
Device: Spinal Sealant — Spinal Sealant System which will be sprayed over the stitches to close the opening in the dura.
  Arms: Spinal Sealant
Procedure: Standard Methods of Closing of the Dura — Standard methods such as the closing of the dura with stitches.
  Arms: Standard Methods

SUMMARY:
1. To evaluate the safety and efficacy of the Spinal Sealant as an adjunct to sutured dural repair compared with standard of care methods (control) to obtain watertight dural closure intraoperatively in patients undergoing spinal surgery.
2. To evaluate the safety and efficacy of the Spinal Sealant as an adjunct to sutured dural repair compared with standard of care methods (control) to obtain watertight dural closure in patients undergoing spinal surgery up to 90 days post-procedure.

DETAILED DESCRIPTION:
The CSF provides a liquid cushion for the brain and spinal cord. The dura holds in the CSF. In order to do spinal surgery, the doctor will cut an opening in the dura. At the end of surgery, the dura must be sealed in order to keep the CSF from leaking out. The doctor will close the dura with stitches and also a piece of tissue taken from another place on your body, to help close the opening. Other standard sealant methods have included the use of Oxicel, Gelfoam, or fibrin glue, but these methods were not designed for closing the dura.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. Your doctor will see you within 30 days before your operation. At this visit, your medical history will be recorded, and you will be asked questions about any other operations you have had in the past. You will have a complete physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight. You will have a sample of your blood (about 2 tablespoons) collected for kidney and liver function tests to make sure they are functioning properly. You will also be asked to fill out 2 questionnaires about your health, daily activities, and back pain. The questionnaires will take about 20 to 30 minutes to complete. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. Participants in one group will receive the Spinal Sealant. You have a 2 out of 3 chance of being randomly assigned to the spinal sealant group. Participants in the other group will receive other standard methods such as the closing of the dura with stitches. However, you will not know which one of the two treatments you receive. Also, (if needed) a piece of your muscle, fat, or other soft tissue may be taken from another place on your body to help seal the opening. Doctors may also use Oxicel, Gelfoam, or fibrin glue to help with the sealing of the dura .

After your already scheduled spinal surgery, your doctor will try to close the opening in the dura, which may be done with stitches alone or, if needed, stitches and a piece of your muscle, fat, or other soft tissue taken from another place on your body. After this try, if there is still some CSF leaking from the dura, you will be assigned to one of the 2 groups for treatment. If you do not have a CSF leak that needs treatment, you will not be able to take part in this study, and you will not have to come back for any study visits.

Participants assigned to the first group will receive treatment with the Spinal Sealant, which will be sprayed over their stitches to close the opening in their dura. The Spinal Sealant is made of 2 plastic-type liquids. When mixed together, a gel is formed that is mostly made up of water. The gel looks and feels sort of like a soft contact lens. After the doctor tries to seal the opening in the dura, the Spinal Sealant is then sprayed over the stitches. It acts like a thin, stretchy covering to help stop the CSF from leaking out through the stitches until the area has properly healed on its own. It is blue-colored, so that the doctor can see where it has been sprayed. Within 1 to 2 months, the gel is naturally broken down by the body and is removed through the urine.

Participants assigned to the second group will be treated with the doctor's choice of other standard treatments to close the opening in their dura. You will not know which group you were assigned to until after the end of your study participation (about 90 days).

While you are still in the hospital (within 7 days after your operation), you will have a physical exam, and your doctor will do a clinical test to check for any CSF leaks. Also, you will have a sample of your blood (about 2 tablespoons) drawn for kidney and liver function tests.

For follow-up, you will be seen by your doctor at about 30 days and again at about 90 days after your operation. It will be very important for you to return to see your doctor at your scheduled follow-up visits, even if you are feeling fine. At the follow-up visits, your doctor will perform a physical exam and check to see how your dura wound is healing and if there is any CSF leakage. You will have a sample of your blood (about 2 tablespoons) collected for kidney and liver function tests. You will also be asked to fill out 2 questionnaires about your health, daily activities, and back pain. The questionnaires will take about 20 to 30 minutes to finish.

Your participation in this study will be over after your 90-day follow-up visit.

THIS IS AN INVESTIGATIONAL STUDY. The Spinal Sealant has been authorized by the FDA for use in research only.

About 158 patients will take part in this multicenter study. Between 15 to 20 participants will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 75 years of age.
2. Patient is scheduled for a spinal procedure that entails a dural incision.
3. Patient requires a procedure involving surgical wound classification Class I/Clean (per CDC criteria).
4. Patient, or authorized representative, has been informed of the nature of the study, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site.
5. Intraoperative Criteria: Presence of non-watertight closure, either spontaneously or upon Valsalva maneuver to 20-25 cm H20 for 5-10 seconds.

Exclusion Criteria:

1. Patient has active spinal and/or systemic infection.
2. Patient will require additional spine surgery within the study time period.
3. Patient has had a previous spinal surgery involving dural exposure and/or entry at the same level(s) as the study procedure.
4. Patient has pre-existing external lumbar CSF drain or internal CSF shunt.
5. Patient is participating in a clinical trial of another investigational device or drug.
6. Patient with creatinine > 2.0 mg/dL.
7. Patient with total bilirubin > 2.5 mg/dL.
8. Pregnant or breast-feeding females or females who wish to become pregnant during the length of study participation.
9. Patient has been treated with chronic steroid therapy unless discontinued more than 6 weeks prior to surgery (standard perioperative steroids are permitted). For purposes of this protocol, chronic steroid therapy is defined as greater than 4 weeks.
10. Patient has documented history of significant coagulopathy with a PTT > 35 sec, PT/ INR >1.2, receiving aspirin, or NSAIDS at the time of surgery. Note: Patients who are receiving cardiovascular prophylaxis are not excluded.
11. Patient is receiving warfarin or heparin at the time of surgery (including analogs).
12. Patient has a diagnosed and documented compromised immune system and/or autoimmune disease.
13. Patient has had chemotherapy treatment within 6 months prior to, or planned during the study (until completion of last follow-up evaluation).
14. Patient has had prior radiation treatment to the surgical site or has planned radiation therapy within 30 days post procedure.
15. Patient has a known malignancy or another condition with prognosis shorter than 6 months.
16. Patients has a documented history of uncontrolled diabetes.
17. The investigator determines that the patient should not be included in the study for reason(s) not already specified.
18. Intraoperative Criteria: Patient requires use of a synthetic or non-autologous duraplasty material.
19. Intraoperative Criteria: Patient has a gap of greater than 2mm remaining after primary dural closure.
20. Patient has undergone laminoplasty decompression.
21. Patient has undergone a Chiari Malformation procedure that does not entail a dural incision at or below the C1 level.
22. Investigator determines that participation in the study may jeopardize the safety or welfare of the patient.
23. Patient has undergone a syringomyelia procedure where the shunt is not placed in the subarachnoid position.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percent (%) success obtaining watertight closure following assigned treatment (Spinal Sealant or control) | Determination in course of surgery with up to 90 day post operative follow-up.
  Percentage (%) success in obtaining a watertight closure following assigned treatment (Spinal Sealant or control) defined as either Success (A watertight closure of the dural repair intra-operatively after assigned treatment, confirmed by Valsalva maneuver at 20-25 cm H2O for 10-15 seconds); or Failure (A non-watertight closure of the dural repair intra-operatively after assigned treatment, confirmed by Valsalva maneuver at 20-25 cm H2O for 10-15 seconds). This will be determined intraoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ian E. McCutcheon, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org